CLINICAL TRIAL: NCT01587222
Title: Midodrine, Octreotide and Albumin: Impact on Renal Function of Patients With Liver Cirrhosis and Renal Failure
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: the sponsor did not provide the treatment
Sponsor: Anna Cruceta (Other)
Responsible Party: Sponsor-Investigator, Anna Cruceta, CTU- Clinical trial unit, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAFRI-II
Record Dates: First submitted 2012-04-27; First posted 2012-04-30 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2015-09

CONDITIONS: Fibrosis; Renal Failure; Hepatorenal Syndrome
MeSH Terms: conditions — Fibrosis; Renal Insufficiency; Hepatorenal Syndrome | interventions — Albumins; Midodrine; Octreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Albumin, Midodrine, Octreotide (Experimental)
  Interventions: Drug: Albumin; Drug: Midodrine; Drug: Octreotide

INTERVENTIONS:
Drug: Albumin — Albumin (20%) 1g/kg iv on day 1 and 80 g every 2 weeks during a period of 12 weeks.
Drug: Midodrine — Oral midodrine 5 mg / 8 hours for 12 weeks. The dose may be increased on day 7 10mg/8h.
  If creatinine does not decrease ≥ 25% and systolic blood pressure is bellow 150 mmHg and diastolic 90 mmHg doses will be changed.
Drug: Octreotide — Octreotide by subcutaneous injection 0.1 mg every 8 hours for 12 weeks. The dose may be increased to 0.2 mg / 8 h on day 7.
  If creatinine does not decrease ≥ 25% and systolic blood pressure is bellow 150 mmHg and diastolic 90 mmHg doses will be changed.

SUMMARY:
The aim of this study is to evaluate the treatment with midodrine, octreotide and albumin during 12 weeks in patients with hepatorenal syndrome. Fifteen patients will be enrolled and followed during 16 weeks. The effects on renal function will be evaluated 12 and 16 weeks after the beginning of the treatment by isotopic evidence and biochemist determinations. Also it will be evaluated arterial pressure and determination of vasoactive hormones (plasma renin, aldosterone and norepinephrine).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80 years
* Cirrhosis of the liver defined by clinical, biochemical or histological
* Functional renal failure with serum creatinine greater than 1.2 mg / dl and less than 2.5 mg / dl.
* That, properly informed, give their consent to participate in the study and undergo tests and examinations that entails
* Women of childbearing potential: pregnancy test negative serum or urine, and acceptance of use of adequate contraception since at least 14 days prior to the first dose of study drug until 14 days after the last dose

Exclusion Criteria:

* Pregnant women, nursing mothers, or those who intend to become pregnant during the study period
* Systolic blood pressure ≥ 150 mmHg and / or diastolic blood pressure ≥ 90 mmHg
* Previous treatment with transjugular intrahepatic portosystemic shunt (TIPS) or surgical portosystemic shunts
* Use of antibiotics in the seven days prior to inclusion in the study except for prophylactic (ie. prophylaxis of spontaneous bacterial peritonitis)
* Cardiac or respiratory failure
* Positive for human immunodeficiency virus
* Urinary retention
* Ischemic heart disease or peripheral vascular disease.
* Narrow Angle Glaucoma
* Cerebrovascular occlusions
* Aortic Aneurysm
* Thyrotoxicosis
* Pheochromocytoma

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-07 (Estimated); Primary Completion 2017-07 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration | 12 weeks
  Change in glomerular filtration rate measured by isotopic tests

SECONDARY OUTCOMES:
Changes in plasma renin activity, plasma aldosterone and norepinephrine | 4, 12 and 16 weeks
Changes in blood pressure measured by Holter | 4, 12 and 16 weeks
Changes in renal function | at 4 weeks after cessation of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic i Provincial de Barcelona, Barcelona, Spain